CLINICAL TRIAL: NCT05942248
Title: The Use of Image-Based Computer Gradings in the Analysis of Acne, Rosacea, Melasma, and Seborrheic Dermatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Codex Labs (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DERM_AI_IMAGES
Record Dates: First submitted 2023-06-14; First posted 2023-07-12 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Acne; Melasma; Rosacea; Seborrheic Dermatitis
Keywords: Artificial Intelligent; Skin
MeSH Terms: conditions — Acne Vulgaris; Melanosis; Rosacea; Dermatitis, Seborrheic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Acne vulgaris (Other): Inflammatory and non-inflammatory lesion counts
  Interventions: Other: No Intervention
- Rosacea (Other): Inflammatory lesion count
  Interventions: Other: No Intervention
- Melasma (Other): Pigment intensity and distribution with use of Melasma Area Severity Index
  Interventions: Other: No Intervention
- Seborrheic Dermatitis (Other): Grading of seborrheic dermatitis with Seborrheic Dermatitis Area Severity Index score
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The study is conducted to determine if image-based computer grading can of acne, melasma, rosacea and seborrheic dermatitis correlate well to expert based clinical severity grading.

DETAILED DESCRIPTION:
The study is conducted to determine if image-based computer grading can of acne, melasma, rosacea and seborrheic dermatitis correlate well to dermatologist based clinical severity grading.

ELIGIBILITY:
Inclusion Criteria:

* Adults with acne, rosacea, melasma or seborrheic dermatitis

Exclusion Criteria:

* Prisoners
* Adults unable to consent
* Artificial facial markings on day of facial photography (such as piercings and tattoos) that may interfere with imaging in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Correlation of image-based grading to clinical gradings for acne | Baseline
  Number of inflammatory and noninflammatory lesions compared to clinical grading
Correlation of image-based grading to clinical gradings for rosacea | Baseline
  Inflammatory lesion count compared to clinical grading
Correlation of image-based grading to clinical gradings for melasma | Baseline
  Melasma area severity index image based grading compared to clinical grading
Correlation of image-based grading to clinical gradings for seborrheic dermatitis | Baseline
  Seborrheic dermatitis area severity index

SECONDARY OUTCOMES:
Sebum excretion rate | Baseline
  Measure of skin sebum via sebumeter

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD, MS, AP, Principal Investigator — Integrative Skin and Research
Locations (1):
- Integrative Skin and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No